CLINICAL TRIAL: NCT02881333
Title: Evaluation of Tools for the Simultaneous Detection of Point and Structural Mutations in Patients With Intellectual Disability
Brief Title: Various Type of Genetic Events in Patients With Intellectual Disability
Acronym: CNV-Seq
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6374
Record Dates: First submitted 2016-08-16; First posted 2016-08-26 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Intellectual Disability
MeSH Terms: conditions — Intellectual Disability | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: Blood samples

SUMMARY:
Currently, for a patient with intellectual disability without a recognizable syndrome (most cases), the way to diagnosis is often long, tedious and expensive because different approaches are used one after the other to identify structural variants (duplications, deletions and other) and point mutations (sequencing of one or more candidate genes). The development of high-throughput sequencing techniques (next generation sequencing: NGS) has drastically increased the detection of point mutations offering the possibility to test a large number of genes simultaneously. NGS also shows a huge potential in detecting structural variants. The objective of this research is to assess the sensitivity of a simultaneous detection of point mutations and structural variants by NGS approaches. This would bring together in a single step the equivalent of performing an array-Comparative genomic hybridization (CGH) analysis plus performing a targeted sequencing of candidate genes. Investigators will compare two approaches for this simultaneous detection: a targeted enrichment of candidate genes coding regions using probes covering these regions associated with a backbone of genomic probes, an approach that could be implemented immediately in diagnostic at the hospital, and a whole genome sequencing (WGS), that is currently a too expensive tool for routine diagnosis but that should be the approach used in the future. Investigators will compare these two approaches to the traditional one: CGH array + WGS. The implementation of a "one step" strategy to detect both types of mutations (punctual and structural) would accelerate and improve the access of patients to a molecular diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with developmental disabilities
* No etiologic diagnosis but suspected genetic cause
* Fragile X syndrome research negative

Exclusion Criteria:

* Children born to consanguineous couples
* Diagnosis already established or suspected
* Identification of an independent etiology

Ages: 3 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with intellectual deficit without diagnosis
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-09 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Detection of mutation from the CGH-array technology on 475 genes | One year

IPD SHARING:
Plan to Share IPD: No